CLINICAL TRIAL: NCT03895528
Title: A Treatment IND (Investigational New Drug) Protocol for EAP (Expanded Access Program) for the Use of Lonafarnib in Patients With Hutchinson-Gilford Progeria Syndrome (HGPS) or Progeroid Laminopathy
Brief Title: Lonafarnib for Patients With Hutchinson-Gilford Progeria Syndrome or Progeroid Laminopathy
Status: Approved for marketing | Type: Expanded Access
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EIG-EAP-LNF-001
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Progeria; HGPS
MeSH Terms: conditions — Progeria | interventions — lonafarnib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Lonafarnib — Farnesyl transferase inhibitor
  Other Names: FTI

SUMMARY:
This treatment IND protocol will allow patients with HGPS and progeroid laminopathies access to lonafarnib, the only compound shown to have an effect on the HGPS disease process resulting in improved outcomes (Gordon et al, 2018). There are no approved treatments for HGPS and progeroid laminopathies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HGPS or progeroid laminopathy by qualified medical doctor (based on common phenotype as described in Gordon 2015 and Merideth 2008). Confirmation with genetic testing is preferred but not required.
* Adequate hepatic function as defined by SGPT (ALT) and SGOT (AST) ≤ 5 times upper limit of normal range for age

Exclusion Criteria:

* Taking medications or foods that are known to be moderate or strong inducers or inhibitors of CYP3A4 or sensitive CYP3A substrates; or if a patient is taking one of these drugs and cannot safely discontinue or take an alternative drug, the dose of the inhibitor/inducer must be adjusted per the treating physician
* Taking digoxin, a P-gp substrate with a narrow therapeutic window.
* Severe renal impairment (GFR < 30 mL/min/1.73m2).
* Uncontrolled infection.
* Presence of any active clinically relevant medical condition that in the opinion of the treating physician would preclude patient from safely participating in the program.
* Pregnant or breast-feeding or plan to become pregnant while on therapy.

Min Age: 12 Months | Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- [Background] Gordon LB, Shappell H, Massaro J, D'Agostino RB Sr, Brazier J, Campbell SE, Kleinman ME, Kieran MW. Association of Lonafarnib Treatment vs No Treatment With Mortality Rate in Patients With Hutchinson-Gilford Progeria Syndrome. JAMA. 2018 Apr 24;319(16):1687-1695. doi: 10.1001/jama.2018.3264. PMID 29710166